CLINICAL TRIAL: NCT06990516
Title: An Open-label, Multi-center Phase Ib/II Clinical Study of the Combination Regimen of SHR - A1811 Injection in the Treatment of Platinum-sensitive Recurrent Ovarian Cancer
Brief Title: SHR - A1811 Injection in the Treatment of Platinum-sensitive Recurrent Ovarian Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Qinglei Gao, Prof., Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-TJ-OVA1811S
Record Dates: First submitted 2025-05-18; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Carboplatin; Oxaliplatin; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-A1811 (Experimental): SHR-A1811: Administered at 3.2 mg/kg, 4 mg/kg, or 4.8 mg/kg intravenously every 3 weeks (Q3W). Carboplatin: Administered at an area under the concentration-time curve (AUC) of 5 mg/mL/min intravenously every 3 weeks (Q3W). Oxaliplatin: Administered at 85 mg/m² intravenously every 3 weeks (Q3W). Bevacizumab: Administered at 15 mg/kg intravenously every 3 weeks (Q3W).
  Treatment duration:
  Platinum - based drugs (carboplatin or oxaliplatin) will be administered for a maximum of 6 cycles or until the occurrence of any event meeting the protocol - defined criteria for treatment discontinuation, whichever occurs first.
  SHR-A1811 and bevacizumab will be continued until the occurrence of any event meeting the protocol - defined criteria for treatment discontinuation.
  Interventions: Drug: SHR-A1811; Drug: Carboplatin; Drug: Oxaliplatin; Drug: Bevacizumab

INTERVENTIONS:
Drug: SHR-A1811 — Dose: 3.2 mg/kg, 4 mg/kg, or 4.8 mg/kg, administered intravenously (IV) every 3 weeks (Q3W).
  Infusion Duration:
  First infusion: 90 ± 10 minutes. Subsequent infusions: May be shortened to approximately 30 minutes (minimum 20 minutes, maximum 60 minutes, including flush phase) if no infusion-related reactions occur after the first dose.
Drug: Carboplatin — Dose: Area Under the Curve (AUC) 5 mg/mL/min, administered IV Q3W.
  Infusion Duration:
  Should be completed within 30-60 minutes (including flush phase).
  Treatment Schedule:
  Up to 6 treatment cycles, with each cycle lasting 3 weeks.
Drug: Oxaliplatin — Dose: 85 mg/m², administered IV Q3W.
  Infusion Duration:
  Should be infused over >120 minutes (including flush phase).
  Treatment Schedule:
  Up to 6 treatment cycles, with each cycle lasting 3 weeks.
Drug: Bevacizumab — Dose: 15 mg/kg, administered IV Q3W.
  Infusion Duration:
  First dose: 90 minutes. Second dose: If the first infusion is well-tolerated, may be shortened to 60 minutes.
  Subsequent doses: If the 60-minute infusion is well-tolerated, all following infusions may be administered over 30 minutes (including flush phase).

SUMMARY:
This study is a multi - center, single - arm, open - label, phase Ib/II clinical trial for dose exploration and efficacy expansion. The aim is to evaluate the tolerability, safety, pharmacokinetic characteristics, and immunogenicity of the combination regimen of SHR - A1811 in the treatment of platinum - sensitive recurrent epithelial ovarian cancer, determine the recommended phase II dose (RP2D) of the combination therapy, and preliminarily assess its efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily joins this study, signs the informed consent form, demonstrates good compliance, and is able to cooperate with follow - up visits.
2. Female, aged 18 - 75 years old (inclusive of 18 and 75 years, calculated from the date of signing the informed consent form).
3. Pathologically diagnosed with epithelial ovarian cancer, fallopian tube cancer, or primary peritoneal cancer (excluding mucinous carcinoma) through tissue or cytology.
4. Has previously received 1 - 3 lines of platinum - containing regimens, and the disease has progressed or recurred (platinum - sensitive recurrence) ≥6 months (183 days) after the end of the last platinum - containing treatment. There must be evidence showing disease progression or recurrence (such as cytology reports of newly - developed ascites or pleural effusion) during or after the last platinum - containing treatment. Solely an elevated CA - 125 level cannot be regarded as evidence of disease progression or recurrence. The combined neoadjuvant and/or adjuvant treatment is counted as one line of treatment. Maintenance treatment is not counted separately. Treatment regimens switched due to reasons other than disease progression (such as toxicity intolerance) are considered part of the same line of treatment and are not counted separately.
5. Has documented mutations in breast cancer susceptibility genes (BRCA 1/2) (germline or somatic) or is homologous recombination deficiency (HRD) positive, and has previously received poly (ADP - ribose) polymerase (PARP) inhibitor treatment.
6. Is able to provide sufficient fresh or archived tumor tissue specimens for the sponsor - designated third - party central laboratory to test the HER2 expression level. The test results do not affect enrollment.
7. Has at least one measurable lesion that meets the RECIST v1.1 criteria (according to the RECIST v1.1 requirements, the long diameter of the measurable lesion on spiral CT scan is ≥10 mm or the short diameter of the enlarged lymph node is ≥15 mm). Lesions that have undergone local treatment can be selected as target lesions if there is clear evidence that they have significantly progressed compared with the post - treatment state.
8. Eastern Cooperative Oncology Group (ECOG) performance status (PS) score: 0 - 1.
9. Expected survival time ≥12 weeks.
10. The functions of important organs meet the following requirements (no blood components or cytokine correction treatments have been used within 14 days before the examination):

    1. Absolute neutrophil count (ANC) ≥1.5×10⁹/L;
    2. Platelet count (PLT) ≥100×10⁹/L;
    3. Hemoglobin (Hb) ≥90 g/L;
    4. Serum albumin (ALB) ≥30 g/L;
    5. Total bilirubin ≤1.5× the upper limit of normal (ULN);
    6. Activated partial thromboplastin time (APTT) ≤1.5×ULN;
    7. International normalized ratio (INR) or prothrombin time (PT) ≤1.5×ULN;
    8. Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≤2.5×ULN (for patients with liver metastases, ALT and/or AST ≤5×ULN);
    9. Serum creatinine (Cr) ≤1.5×ULN or creatinine clearance rate (Clcr) ≥50 mL/min (calculated according to the Cockcroft - Gault formula);
    10. QTc ≤470 msec;
    11. Left ventricular ejection fraction (LVEF) ≥50%, and the cardiac function test results should be completed within 28 days before the first administration of the drug;
    12. Urine protein <2+. If urine protein ≥2+, the 24 - hour urine protein quantification must show that the protein is <1 g.
11. Female subjects of childbearing potential must have a negative serum human chorionic gonadotropin (HCG) test within 7 days before the first administration of the drug, and must not be breastfeeding. Female subjects of childbearing potential must agree to comply with contraceptive requirements from the date of signing the informed consent form until 7 months after the last administration of the investigational drug.

Exclusion Criteria:

1. Subjects with untreated or active central nervous system (CNS) tumor metastases. Subjects with a history of leptomeningeal metastasis or current leptomeningeal metastasis. Subjects whose CNS tumor metastases have undergone adequate local treatment (surgery or radiotherapy), do not require hormone therapy, have neurologically returned to baseline (except for residual signs or symptoms related to CNS treatment), and have been stable for ≥4 weeks can be enrolled.
2. Subjects with a history of or currently having other malignancies, except for cured basal cell carcinoma of the skin, cervical intraepithelial neoplasia, ductal carcinoma in situ of the breast, papillary thyroid carcinoma, and other malignancies that have been adequately treated and cured for ≥3 years before randomization with evidence proving no recurrence or metastasis.
3. Subjects with symptomatic, poorly controlled, or moderate - to - severe pleural effusion, pericardial effusion, or ascites; subjects who have undergone effusion drainage (except diagnostic thoracentesis) can be enrolled if they have been stable for at least 2 weeks after drainage (local treatment within the serous cavity according to routine diagnosis and treatment is allowed before signing the informed consent form).
4. Subjects with a history of interstitial pneumonia/interstitial lung disease or non - infectious pneumonia (such as radiation pneumonitis, etc.) that required steroid treatment; subjects with current or suspected interstitial pneumonia/interstitial lung disease, non - infectious pneumonia, or other active pneumonias; subjects who had severe asthma, severe chronic obstructive pulmonary disease (COPD), or restrictive lung disease and other lung damages within 6 months before the first administration of the drug.
5. Subjects with active pulmonary tuberculosis; subjects who have undergone regular and adequate treatment before the first administration of the drug and have stopped anti - tuberculosis treatment for ≥3 months can be enrolled.
6. Subjects with hypertension that cannot be well - controlled by antihypertensive drugs (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg, based on the average value of blood pressure readings obtained from at least 2 measurements, and the above parameters can be achieved through antihypertensive treatment), and subjects who have had hypertensive crisis or hypertensive encephalopathy in the past.
7. Subjects with uncontrolled or severe cardiovascular diseases, such as unstable angina, symptomatic congestive heart failure (New York Heart Association [NYHA] class II - IV), myocardial infarction within 6 months before the first administration of the drug, or unstable angina or unstable arrhythmia within 1 month before the first administration of the drug.
8. Subjects who have had arterial or venous thrombotic events within 6 months before the first administration of the drug, including but not limited to cerebrovascular accidents, deep vein thrombosis, and pulmonary embolism; subjects with intramuscular vein thrombosis or catheter - related thrombosis of the infusion port before the first administration of the drug can be included if the investigator judges there is no risk.
9. Subjects who have had NCI - CTCAE v5.0 - graded ≥Grade 2 bleeding events within 1 month before the first administration of the drug, including but not limited to hemoptysis (a single episode of hemoptysis volume ≥2 mL), vaginal bleeding, gastrointestinal bleeding; or subjects with radiation enteritis accompanied by bleeding symptoms during the screening period; subjects with positive fecal occult blood retest at baseline and judged by the investigator to have a bleeding risk cannot be enrolled.

   Note: Transient bleeding caused by iatrogenic operations is excluded.
10. Subjects with known hereditary or acquired bleeding (such as coagulation disorders, hemophilia) or thrombotic tendency; subjects who have used anti - platelet drugs such as aspirin (>325 mg/d), clopidogrel, ticagrelor within 14 days before the first administration of the drug; subjects who have used anticoagulant therapy for therapeutic purposes within 2 weeks before the first administration of the drug [low - dose aspirin and low - molecular - weight heparin (such as enoxaparin sodium ≤40 mg/d) for preventive use are allowed].
11. Subjects who have had gastrointestinal perforation or fistula, tracheal fistula, urethral fistula, or abdominal abscess within 3 months before the first administration of the drug or are expected to have them in the near future; subjects who have undergone artificial fistulization or ureteral stent placement and are considered stable by the investigator after evaluation can be enrolled.
12. Subjects with gastrointestinal obstruction or symptoms and signs of gastrointestinal obstruction within 6 months before the first administration of the drug, but subjects who have undergone surgical treatment and the obstruction has been completely relieved can be screened; subjects who have previously undergone intestinal stent implantation and the intestinal stent has not been removed until the screening period.
13. Subjects who have had severe infections within 1 month before the first administration of the drug, including but not limited to infection complications requiring hospitalization, bacteremia, severe pneumonia, etc.; subjects with any active infections requiring intravenous systemic treatment, or subjects who have unexplained fever >38.5°C during the screening period or before the first administration of the drug.
14. Subjects with a history of immunodeficiency, including positive HIV test results, other acquired or congenital immunodeficiency diseases, or a history of organ transplantation; subjects with active hepatitis (for hepatitis B: HBsAg positive and HBV DNA detection value ≥500 IU/mL (if the research center only has copy/mL as the detection unit, subjects with ≥2500 copy/mL are not eligible), or active hepatitis C (defined as positive HCV - Ab test result during the screening period and positive HCV - RNA)).
15. Subjects who underwent surgery (except diagnostic surgery), radical radiotherapy, chemotherapy, large - molecule targeted therapy, or anti - tumor immunotherapy, and the time from the completion of treatment (last medication) to the first administration of the drug is less than 4 weeks; subjects who used small - molecule targeted drugs (including other investigational oral targeted drugs) and the time from the last medication to the first administration of the drug is less than 5 half - lives or 4 weeks (whichever is shorter); subjects who underwent palliative radiotherapy or local treatment, and the time from the completion of treatment to the first administration of the drug is less than 2 weeks.
16. Subjects who have previously received anti - HER2 treatment (such as HER2 ADC), or antibody - drug conjugates containing topoisomerase I inhibitors, or topoisomerase I inhibitor treatment (such as irinotecan, topotecan).
17. Subjects who may receive other systemic anti - tumor treatments during the study or plan to undergo secondary cytoreductive surgery.
18. According to the NCI - CTCAE v5.0 grading system, subjects whose toxicity caused by previous anti - tumor treatment has not recovered to ≤Grade 1 (except for decreased lymphocyte count, alopecia, fatigue, and laboratory indicators mentioned in the inclusion criteria; some tolerable chronic Grade 2 toxicities can be excluded after consultation between the investigator and the sponsor).
19. Subjects who are known to be allergic to any component of the SHR - A1811 product (antibody - conjugated toxin, antibody, toxin SHR169265) or to any platinum - containing drug.
20. In the opinion of the investigator, subjects with other factors that may affect the study results or lead to the premature termination of this study, such as alcoholism, drug abuse, drug addiction, criminal detention, etc., as well as other serious diseases (including mental illnesses) requiring concomitant treatment, severe laboratory abnormalities, and other any conditions that may increase the risk of participating in the study, interfere with the study results, or make the subject unsuitable for this study.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Ovarian cancer patients
Enrollment: 90 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2030-06-01 (Estimated); Study Completion 2035-06-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR): | 5 Years after treatment.
  Defined as the proportion of subjects who achieve a Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR) as assessed by the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1). For responses categorized as CR or PR, confirmation is required through a subsequent evaluation performed no less than 4 weeks (≥28 days) after the initial assessment.

SECONDARY OUTCOMES:
Duration of Response (DoR) | 5 Years after treatment.
  Defined as the time from the first date a subject is assessed as having a confirmed Complete Response (CR) or Partial Response (PR) to the first date of either Progressive Disease (PD) or death due to any cause, whichever occurs first.
Disease Control Rate (DCR) | 5 Years after treatment.
  Defined as the proportion of subjects with a Best Overall Response (BOR) of Complete Response (CR), Partial Response (PR), or Stable Disease (SD) as assessed by the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).
Response Rate (RR) | 5 Years after treatment.
  Defined as the proportion of subjects with an overall response assessed as either a response according to the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) or a response according to the Gynecologic Cancer InterGroup (GCIG) CA - 125 criteria.
CA - 125 Response Rate (CA - 125 RR) | 5 Years after treatment.
  Defined as the proportion of subjects with a response evaluated according to the Gynecologic Cancer InterGroup (GCIG) CA - 125 criteria.
Progression Free Survival | 5 Years after treatment.
  Progression - Free Survival (PFS) as assessed by the Independent Radiological Review Committee (IRC) based on the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1). It is defined as the time from the randomization date of the subject to the first date of documented radiological tumor progression or the date of death due to any cause, whichever occurs first.
Overall Survival (OS) | 5 Years after treatment.
  Defined as the time from the randomization date to death due to any cause in subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Qinglei Gao, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
Contact Prof. Gao for primary data.